CLINICAL TRIAL: NCT02217345
Title: Growth Hormone and Intrahepatic Lipid Content in Patients With Nonalcoholic Fatty Liver Disease
Acronym: NAFLD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Karen Klahr Miller, MD, Neuroendocrine Unit Chief, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2014P001680
Record Dates: First submitted 2014-07-15; First posted 2014-08-15 (Estimated); Results first posted 2022-11-22 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-10

CONDITIONS: Nonalcoholic Fatty Liver Disease (NAFLD)
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Growth Hormone; Human Growth Hormone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Growth hormone (Experimental): Growth hormone (somatropin) administered by daily injection at starting dose of 0.3 mg daily for women and 0.2 mg daily for men, with dose titration for goal IGF-1 in the upper quartile of normal for age.
  Interventions: Drug: Growth hormone
- Placebo (Placebo Comparator): Placebo will be administered by daily injection in this double blind study design. Sham dosing will be performed to maintain blinding.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Growth hormone — growth hormone, Genotropin (Pfizer)
  Other Names: Genotropin (Pfizer Inc.)
  Arms: Growth hormone
Drug: Placebo — placebo with identical drug pen delivery device and packaging as Genotropin (Pfizer)
  Arms: Placebo

SUMMARY:
Nonalcoholic fatty liver disease (NAFLD), fatty infiltration of the liver in the absence of alcohol use, is an increasingly recognized complication of obesity, with prevalence estimates of about 30% of individuals in the United States. A subset of these will develop progressive disease in the form of nonalcoholic steatohepatitis (NASH), which can progress to cirrhosis and liver failure. NAFLD is expected to be the most common indication for liver transplantation by the year 2020. We hypothesize that growth hormone (GH) replacement will decrease intrahepatic lipid accumulation as quantified by 1H magnetic resonance spectroscopy (1H-MRS).

ELIGIBILITY:
Inclusion Criteria:

1. Ages 18 - 65 yr
2. NAFLD defined as demonstration of hepatic steatosis by imaging or biopsy in absence of significant alcohol consumption and other causes of hepatic steatosis. If liver imaging or biopsy has not been performed clinically, liver ultrasound will be performed as part of the screening visit.

Exclusion Criteria:

1. Serum creatinine > 2 times the upper limit of normal
2. History of cancer, except for non-melanoma skin cancers
3. Active carpel tunnel syndrome
4. Diabetes mellitus, defined as a hemoglobin A1C >6.5 or use of any medications prescribed to treat hyperglycemia. The exception is that the use of metformin is acceptable in patients whose HbA1c has been =<6.0 on two visits and whose weight has remained stable for six months.
5. Contraindications to magnetic resonance imaging (MRI).
6. Pregnancy or desire to become pregnant. Participants of reproductive age must agree to use contraception.
7. Breastfeeding
8. Aspartate and aminotransferase levels >10x upper limit of normal

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2017-06-02 (Actual); Primary Completion 2021-08-10 (Actual); Study Completion 2021-09-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen K Miller, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited through hospital-wide and community advertisements between 2017-2021. Recruitment techniques included posting advertisements on the internet (i.e. Craigslist and Facebook) and on the Massachusetts General Hospital's clinical trial recruitment website.
Pre-assignment Details: Of the 131 people who signed a consent form, 78 were unable to participate due to various reasons including meeting ineligibility criteria. The 53 subjects who remained were randomized to one of two arms. One subject discontinued after randomization but before any baseline procedures were completed, leaving 52 subjects with available baseline data.
Groups:
- Growth Hormone: Growth Hormone (GH) is Genotropin, provided by Pfizer Inc. It is a self-administered sub-cutaneous daily injection using an injection pen device. It was administered for 6 months. The dose was titrated based on IGF-1 hormone levels with the goal of maintaining an IGF-1 level in the upper-quartile of the normal range.
- Placebo: Placebo was provided by Pfizer Inc. It appeared identical to active growth hormone and was administered in the same manner; self-administered sub-cutaneous daily for 6 months using an injection pen device. Dose was titrated in a way to maintain the double-blind.
Period: Overall Study
Arm/Group | Growth Hormone | Placebo
Started | 27 | 26
Baseline Data Available | 26 | 26
Completed | 20 | 21
Not Completed | 7 | 5
Not completed — Lost to Follow-up | 2 | 1
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Adverse Event | 2 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Population: One subject discontinued after randomization but before any baseline procedures were completed, leaving 52 subjects with available baseline data.
Groups:
- Total: Total of all reporting groups
Arm/Group | Growth Hormone | Placebo | Total
Number analyzed (Participants) | 26 | 26 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 26 | 51
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (12) | 46 (12) | 46 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 26
  Male | 13 | 13 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 26 | 24 | 50
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 2 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 19 | 20 | 39
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 26 | 26 | 52

OUTCOME MEASURES:

1. Primary Outcome: Change in Intrahepatic Lipid Content Between Baseline and 6 Months as Measured by 1H-magnetic Resonance Spectroscopy (1H-MRS). Endpoints Were Assessed at Baseline and 6 Months.
Description: Change in Intrahepatic lipid content by 1H-MRS over 6 months in the GH vs placebo group
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: percent liver fat
Arm/Group | Growth Hormone | Placebo
Number analyzed (Participants) | 20 | 21
percent liver fat | -5.2 (10.5) | 3.8 (6.9)

2. Secondary Outcome: Change in Serum High Sensitivity C-reactive Protein (hsCRP) Between Baseline and 6 Months.
Description: Change in serum high sensitivity C-reactive protein (hsCRP) (mg/L) between baseline and 6 months.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Growth Hormone | Placebo
Number analyzed (Participants) | 20 | 21
mg/L | -0.8 (0.9) | 0.3 (1.7)

ADVERSE EVENTS:
Time Frame: 6 months
Description: GH is FDA approved. Adverse events were defined by the clinicaltrials.gov definitions and categorized as "expected" and "unexpected" based on the medication package insert.
  GH group: 27 randomized and 3 pre-drug discontinuations = 24 at risk Placebo group: 26 randomized and 1 pre-drug discontinuation = 25 at risk
  # of events = # of subjects that experienced the side effect at any point during the study.
Arm/Group | Growth Hormone | Placebo
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/25
Serious Adverse Events (participants affected / at risk) | 1/24 | 0/25
Other Adverse Events (participants affected / at risk) | 15/24 | 11/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Growth Hormone (N=24) | Placebo (N=25)
Unrelated surgical procedure (Surgical and medical procedures) | 1 (1) | 0 (0) — unrelated SAE
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Growth Hormone (N=24) | Placebo (N=25)
Edema (Blood and lymphatic system disorders) | 5 (5) | 0 (0) — (swelling) in the hands and/or feet
Headache (General disorders) | 3 (3) | 4 (4)
Carpal Tunnel Syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint Pain or Stiffness (Musculoskeletal and connective tissue disorders) | 4 (4) | 6 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Numbness or tingling (Nervous system disorders) | 3 (3) | 2 (2)
Injection site discomfort or bruising (Skin and subcutaneous tissue disorders) | 4 (4) | 5 (5)
Allergic Reaction (Immune system disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
We cannot extrapolate efficacy and safety to patients with diabetes mellitus.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-02-17): https://cdn.clinicaltrials.gov/large-docs/45/NCT02217345/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-17): https://cdn.clinicaltrials.gov/large-docs/45/NCT02217345/SAP_001.pdf